CLINICAL TRIAL: NCT00186173
Title: Sports to Prevent Obesity: Feasibility and Pilot RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Association of American Medical Colleges (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MM-0851-05/05; SPO#31174
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
Keywords: Obesity; Physical activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- After school sports (Experimental): After school team sports intervention designed specifically for overweight and obese children
  Interventions: Behavioral: After school sports program
- After school health education (Active Comparator): After school heath and nutrition education program
  Interventions: Behavioral: After school health education

INTERVENTIONS:
Behavioral: After school sports program — After school team sports intervention designed specifically for overweight and obese children
  Arms: After school sports
Behavioral: After school health education — After school health and nutrition education program
  Arms: After school health education

SUMMARY:
The purpose of this study is to learn whether overweight children who participate in an after school sports program improve their health as much as overweight children in a more traditional health education program.

DETAILED DESCRIPTION:
After school sports programs may be generalizable, motivating and cost-efficient interventions for long-term weight control among at-risk and overweight children. The infrastructure needed to provide such programs already exists in most communities. In contrast, more traditional, medically- and behaviorally-oriented treatment programs are expensive, generally not very effective, often inconvenient, and not available in most communities. While children involved in team sports tend to be more physically fit than their uninvolved peers, team sports has not yet been tested as a method to increase involvement of at-risk and overweight children in regular physical activity. As an added bonus, these sports programs can displace typical after school television viewing and snacking. Team sports is a potentially innovative and high impact approach for intervening with at-risk and overweight children, as it may provide an opportunity to reduce weight gain while increasing social interaction and self-esteem. If our proposed research finds that team sports are an efficacious intervention for reducing weight gain among low-income at-risk and overweight children, it is an intervention approach that could be rapidly diffused and tested for effectiveness. The policy implications of these findings would be great, encouraging expanded access to team sports programs to a population that has not been previously targeted or included.

We propose a two-phase project in East Palo Alto, California, a low-income, primarily Latino, African-American and Pacific Islander community. The first phase will be a 3-month feasibility trial of an after school team sports program for overweight children to examine several theory-driven approaches to program design and implementation, including assessments of liking and participation and barriers and facilitators of participation. The second phase will be a 6-month randomized controlled pilot trial (RCT) comparing weight changes among overweight children randomized to participate in the after school team sports program versus a traditional weight control/health education program.

ELIGIBILITY:
Inclusion Criteria:

* In 4th or 5th grade of a participating school at time of enrollment
* BMI greater than or equal to the 85th percentile on the 2000 CDC growth charts
* Medical clearance obtained from primary care provider

Exclusion Criteria:

Our goal is to be inclusive as possible, however, children will not be eligible to participate if they:

* have a condition that limits their participation in physical activity enough that they are not able to participate in Physical Education at school (e.g. significant structural heart disease)
* are pregnant
* have been diagnosed with a chronic illness that affects their growth and/or weight (e.g., type 1 diabetes, hypothyroidism, inflammatory bowel disease)
* have taken systemic steroids (oral, intravenous, or intramuscular) for a period of more than 21 days in the past year
* are taking other medications potentially affecting their growth and/or weight (e.g. methylphenidate HCL)
* are unable to complete the informed consent process

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-11; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Body mass index | Baseline, 3 and 6 months

SECONDARY OUTCOMES:
Waist circumference | Baseline, 3 and 6 months
Triceps skinfold thickness | baseline, 3 and 6 months
Resting heart rate | baseline, 3 and 6 months
Physical activity monitoring | baseline, 3 and 6 months
Sedentary behaviors | baseline, 3 and 6 months
Psychosocial measures | baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Robinson, MD, MPH, Principal Investigator — Stanford University; Dana L Weintraub, MD, Study Director — Stanford University

REFERENCES:
- [Result] Weintraub DL, Tirumalai EC, Haydel KF, Fujimoto M, Fulton JE, Robinson TN. Team sports for overweight children: the Stanford Sports to Prevent Obesity Randomized Trial (SPORT). Arch Pediatr Adolesc Med. 2008 Mar;162(3):232-7. doi: 10.1001/archpediatrics.2007.43. PMID 18316660